CLINICAL TRIAL: NCT03523754
Title: Intravaginal Isosorbide Mononitrate in Addition to Misoprostol Versus Misoprostol Only for Induction of Labor: A Randomized Controlled Trial
Brief Title: Intravaginal Isosorbide Mononitrate in Addition to Misoprostol Versus Misoprostol Only for Induction of Labor
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dina Yahia Mansour (Other)
Responsible Party: Sponsor-Investigator, Dina Yahia Mansour, Lecturer of Obstetrics & Gynecology, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Vaginal nitric oxide donor
Record Dates: First submitted 2018-02-13; First posted 2018-05-14 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Induction of Labor
Keywords: Induction of labor; isosorbide mononitrate; misoprostol
MeSH Terms: interventions — isosorbide-5-mononitrate; Misoprostol

STUDY DESIGN:
Intervention Model Description: * Primigravida.
  * From 20 to 30 years old.
  * Singleton term (between 40 to 42 weeks of gestation).
  * Good general condition with straightforward enthusiasm for the trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Misoprostol only (Other): This group will receive Intravaginal Misoprostol only.
  Interventions: Drug: Isosorbide Mononitrate 40 MG to study group
- Isosorbide Mononitrate & Misoprostol (Other): This group will reveive intravaginal Isosorbide Mononitrate & Misoprostol.
  Interventions: Drug: Isosorbide Mononitrate 40 MG to study group

INTERVENTIONS:
Drug: Isosorbide Mononitrate 40 MG to study group — Isosorbide Mononitrate will be added to Misoprostol, to determine their combined effect on cervical ripening & induction of labor in study group
  Other Names: Misoprostol 25Mcg

SUMMARY:
Evaluation of safety & efficacy of nitric oxide donors such as intravaginal isosorbide mononitrate in addition to misoprostol Versus misoprostol only for the whole process of induction of labor.

DETAILED DESCRIPTION:
* Type of Study: Randomised controlled clinical trial.
* Study Setting: This study will be conducted at Ain Shams University's Emergency department of the Maternal Hospital.
* Study Period: From January 2018 to June 2018 (6 months)
* Randomization: Will be done using computer generated randomization sheet using MedCalc© version 13. ( Appendix 1)
* Allocation and concealment: Fifty opaque envelops will be numbered serially and in each envelope the corresponding letter which denotes the allocated group will be put according to randomization table. Then all envelopes will be closed and put in one box. When the first patient arrives, the first envelope will be opened and the patient will be allocated according to the letter inside.
* Study Population: Fifty pregnant women.

  * Inclusion Criteria:

    * Primigravida.
    * From 20 to 30 years old.
    * Singleton term (between 40 to 42 weeks of gestation).
    * Good general condition with straightforward enthusiasm for the trial.
  * Exclusion Criteria:

    * IUGR.
    * Rupture of membranes.
    * Favorable cervix (Bishop score : '8' or more)
    * Cephalopelvic disproportion,fetal malpresentation.
    * Antepartum hemorrhage, any abnormal placentation such as placenta previa, morbidly adherent placenta.
    * Uterine fibroid.
    * Previous uterine major surgery such as : myomectomy.
    * Any medical disorder such as : gestational diabetes, diabetes mellitus, hypertension, preeclampsia, coagulation disorders, renal and hepatic dysfunction.
* Sampling Method: Convenience sampling.
* Sample Size: Fifty women.
* Sample Justification: Using data from previous study by Abdellah et al. 2010, which compared isosorbide mononitrate and misoprostol versus misprostol only. Misoprostol only group induction to delivery interval was 23 hours while in the isosorbide mononitrate and misorprostol group it was 19.6 hours. We will use sample size of 25 women in each of the two groups to achieve 91% power to detect statistical difference of atleast 3.4 hours. With estimated group standard deviations of 4.0 and 2.6 and with a significance level (alpha) of 0.05 using Mann-Whitney test; the sample size of 50 women as stated before is satisfactory to detect difference between initial dose to delivery.
* Ethical Considerations: An informed consent will be taken from all participants, it will be in Arabic language and confirmed by date & time. No harm will be inflicted & no benefit will be deprived in this study.
* Study Procedures:

  * Fifty Primigravida women will be recruited according to inclusion and exclusion criteria.
  * History taking.
  * Physical examination.
  * Ultrasound: for placental localization excluding abnormal localization, exclude Fetal IUGR, oligohydraminos, polyhydraminos, fibroids.
  * Laboratory investigations: CBC (complete blood count) , Coagulation Profile, Liver function test, Kidney function test, ABO Rhesus D (RhD).
  * Counseling of the patient about isosorbide mononitrate and misoprostol.
  * Recruited patients will fill a written consent.
  * Two types of envelopes will be available, one with misoprostol & placebo, other will contain misoprostol & isosorbide mononitrate which will be given by vaginal route.
  * Patient will choose an envelope from the previous 2 types.
  * 2 groups will be formed; group 1 will take both misoprostol & isosorbide mononitrate, group 2 will take Misoprostol only. Group 1 will take intial dose of 40mg isosorbide mononitrate (Mono-Mak) in the posterior vaginal fornix which will not be repeated; followed by intravaginal 25mcg of misoprostol (Vagiprost), misoprostol will be repeated every 6 hours for maximum of 5 doses (i.e. 125mcg), (FIGO recommendation for misoprostol regimen 2017 & WHO recommendations for induction of labour 2011). Misoprostol will be stopped when labour is established defined by 3 contractions every 10 minuites, each contraction of 30 seconds duration, with amplitude of 40 mmHg or if 6 hours passed after the last misoprostol dose and labour is not established as defined before with unfavorable cervix defined by bishop score of 6 or less, cesarean delivery will be performed. Group 2 will take only misoprostol with same scheme for misoprostol as before in group 1.
  * Induction of labor process will take place, during which:

    * Maternal blood pressure & pulse will be assessed every 30 minutes for the first 2 hours then hourly after that; temperature will be assessed every 4 hours.
    * Fetal auscultation will be carried out every 15 minutes in 1st stage of labor, every 5 minutes in 2nd stage of labor after uterine contraction for at least 1 minuite.
    * CTG will be performed every 2 hours or if there are concerns during fetal ausculatation. Continuous CTG maybe continued upon maternal request or if there are high risk factors such as contractions that last longer than 60 seconds(hypertonus) or more than 5 contractions in 10 minutes(tachysystole), Oxytocin use.
* Study Interventions: Cesarean Delivery will be performed in the following circumstances:

  * if Induction of labor failure is established defined by unfavorable cervix after 6 hours from the last dose of 5 doses of Misoprostol each is 25 mcg (maximum dose of 125mcg)
  * If management of protraction & arrest disorders failed.
  * If CTG monitoring was classified as pathological and conservative management failed; or if CTG monitoring warned the need for urgent intervention.
* Statistical Analysis: Descriptive statistics for measured variables will be expressed as range mean and standard deviation (for metric data); range, median and interquartile range (for discrete data); and number and proportion (for categorical data). Demographic data and primary and secondary outcomes of all women will be compared using t-test (for quantitative parametric measures), Mann-Whitney's U-test (for quantitative non-parametric measures) and chi squared and Fisher's Exact tests (for categorical measures). Pearson's correlation coefficient (for metric variables) and Spearman's correlation coefficient (for rank variables) will be used to estimate association between variables.
* Statistical Package: Data will be collected, edited and entered into suitable software for data entry & analysis such as 'SPSS version 20'.

ELIGIBILITY:
Inclusion Criteria:

* Primigravida.
* From 20 to 30 years old.
* Singleton term (between 40 to 42 weeks of gestation).
* Good general condition with straightforward enthusiasm for the trial.

Exclusion Criteria:

* IUGR.
* Rupture of membranes.
* Favorable cervix (Bishop score : '8' or more)
* Cephalopelvic disproportion,fetal malpresentation.
* Antepartum hemorrhage, any abnormal placentation such as placenta previa, accreta, increta and percreta
* Uterine fibroid.
* Previous uterine major surgery such as : myomectomy, uterine repair caused by trauma and metroplasty for Mullerian anomalies.
* Any medical disorder such as : gestational diabetes, diabetes mellitus, hypertension, preeclampsia, renal & hepatic dysfunction, coagulation disorders.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women only.
Enrollment: 50 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-10-01 (Estimated); Study Completion 2018-11-30 (Estimated)

PRIMARY OUTCOMES:
Decrease interval between drug use to delivery | 6 months
  Adding Isosorbide Mononitrate to Misoprostol will decrease time required for induction of labor.

CONTACTS AND LOCATIONS:
Overall Officials: Hesham M. Harb, MD, Principal Investigator — Professor of Obstetrics & Gynecology; Dina Y. Mansour, MD, Principal Investigator — Lecturer of Obstetrics & Gynecology; Yahia M. A. Mohamed ELBoukhary A.A., M.B.B.Ch, Principal Investigator — Msc Student, Resident of Obstetrics & Gynecology
Locations (1):
- Department of Obs & Gyn,Faculty of Medicine, Ain shams University., Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
We will see if the study may add new to the scientific society or no, if the study is done, completed in a good environment and we are convinced that it may provide new information to others, we will share it.